CLINICAL TRIAL: NCT06436521
Title: The Efficacy of Online Brief Positive Cognitive Behavior Therapy Compared to Traditional Cognitive Behavior Therapy on Improving Well-Being and Goal Attainment in Young Adults
Brief Title: The Efficacy of Online Brief Positive Cognitive Behavior Therapy Compared to Traditional Cognitive Behavior Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Comsa Loana, Principal Investigator, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MDStudy
Record Dates: First submitted 2024-03-22; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-03

CONDITIONS: Emotional Distress; Well-Being, Psychological; Performance
Keywords: Solution-focused; Problem-solving; Positive CBT; Traditional CBT; Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one approach: Positive CBT or Traditional CBT, through simple randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive CBT (P-CBT) (Experimental): Participants received P-CBT intervention after a standard protocol. The intervention used Solution-focused questioning.
  Interventions: Behavioral: Positive Cognitive Behavioral Therapy
- Traditional CBT (T-CBT) (Experimental): Participants received T-CBT intervention after a standard protocol. The intervention used Problem-solving questioning.
  Interventions: Behavioral: Traditional Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Positive Cognitive Behavioral Therapy — Positive CBT integrates brief Solution-Focused Brief Therapy with Positive Psychology techniques, within a cognitive-behavioral framework. It is considered a competency and strengths-based model.
  Arms: Positive CBT (P-CBT)
Behavioral: Traditional Cognitive Behavioral Therapy — Traditional cognitive behavioral therapy is a form of psychological treatment that emphasizes that psychological problems are based on faulty or unhelpful ways of thinking and the focus is to change thinking patterns.
  Arms: Traditional CBT (T-CBT)

SUMMARY:
Positive Cognitive Behavioral Therapy (P-CBT) has emerged as the fourth Cognitive Behavioral Therapy waive, based on critiques brought to Cognitive Behavioral Therapy for being grounded in the deficit-based medical model. The study aim to identify which of the two Cognitive Behavioral Therapy approaches, Positive or Traditional, is more effective in a brief format in terms of improving emotional state, attaining goals, and changing attitudes in young adults.

DETAILED DESCRIPTION:
This study is a randomized controlled trial that aims to explore the effectiveness of two Cognitive Behavioral approaches: Positive and Traditional, in terms of improving emotional state, attaining goals, and changing attitudes in young adults. Thirty-eight participants divided into two groups, received four therapy sessions for four weeks. The outcomes were measured four times: pre-, mid- (after two sessions), post-intervention (after four sessions), and at two-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Students in the master's program in psychology

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Distress | Baseline, pre-intervention; in the middle of intervention, after 2 sessions (2 weeks); immediately after the intervention (4 weeks); 2 month.
  The level of negative emotions, measured with Profile of Affective Distress plus. The items are ranked with a 5-point Likert scale. Higher scores mean a worse outcome.
Positive Emotions | Baseline, pre-intervention; in the middle of intervention, after 2 sessions (2 weeks); immediately after the intervention (4 weeks); 2 month.
  The level of positive emotions, measured with Profile of Affective Distress plus; The items are ranked with a 5-point Likert scale.Higher scores mean a better outcome.
Performance | Baseline, pre-intervention; in the middle of intervention, after 2 sessions (2 weeks); immediately after the intervention (4 weeks); 2 months.
  Performance was measured using a Visual Analogue Scale -type item. The outcome had a one-item ranging from 1 to 10. Participants had to assess the statement: - How close are you to solving the problem/attaining your goal? Higher scores mean a better outcome.
Attitude towards problems | Baseline, pre-intervention; in the middle of intervention, after 2 sessions (2 weeks); immediately after the intervention (4 weeks); 2 months.
  Measured with Solution Focused Inventory; The items are ranked with a 6-point Likert scale. Higher scores mean a better outcome.
Attitude towards goals | Baseline, pre-intervention; in the middle of intervention, after 2 sessions (2 weeks); immediately after the intervention (4 weeks); 2 months.
  Measured with Solution Focused Inventory; The items are ranked with a 6-point Likert scale. Higher scores mean a better outcome.
Attitude towards resources | Baseline, pre-intervention; in the middle of intervention, after 2 sessions (2 weeks); immediately after the intervention (4 weeks); 2 months.
  Measured with Solution Focused Inventory; The items are ranked with a 6-point Likert scale. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Loana T Comsa, Ph.D., Principal Investigator — Babes-Bolyai University Cluj-Napoca
Locations (1):
- Departement of Clinical Psychology and and Psychotherapy, Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bannink, F. (2012). Practicing positive CBT: From reducing distress to building success. John Wiley & Sons https://doi.org/10.1002/9781118328941
- [Background] Bannink, F., & Geschwind, N. (2021). , Positive CBT: Individual and Group Treatment Protocols for Positive Cognitive Behavioral Therapy. In Positive CBT: Individual and Group Treatment Protocols for Positive Cognitive Behavioral Therapy. https://doi.org/10.1027/00578-000
- [Background] Bhattacharya S, Goicoechea C, Heshmati S, Carpenter JK, Hofmann SG. Efficacy of Cognitive Behavioral Therapy for Anxiety-Related Disorders: A Meta-Analysis of Recent Literature. Curr Psychiatry Rep. 2023 Jan;25(1):19-30. doi: 10.1007/s11920-022-01402-8. Epub 2022 Dec 19. PMID 36534317
- [Background] Braunstein, K., & Grant, A. M. (2016). Approaching solutions or avoiding problems? The differential effects of approach and avoidance goals with solution-focused and problem-focused coaching questions. Coaching, 9(2). https://doi.org/10.1080/17521882.2016.1186705
- [Background] Cohen, J. (1988a). Statistical power analysis for the behavioral sciences (2nd ed.). Hillsdale, NJ: Lawrence Erlbaum Associates.
- [Background] Cuijpers P, Miguel C, Harrer M, Plessen CY, Ciharova M, Ebert D, Karyotaki E. Cognitive behavior therapy vs. control conditions, other psychotherapies, pharmacotherapies and combined treatment for depression: a comprehensive meta-analysis including 409 trials with 52,702 patients. World Psychiatry. 2023 Feb;22(1):105-115. doi: 10.1002/wps.21069. PMID 36640411
- [Background] de Boer AG, van Lanschot JJ, Stalmeier PF, van Sandick JW, Hulscher JB, de Haes JC, Sprangers MA. Is a single-item visual analogue scale as valid, reliable and responsive as multi-item scales in measuring quality of life? Qual Life Res. 2004 Mar;13(2):311-20. doi: 10.1023/B:QURE.0000018499.64574.1f. PMID 15085903
- [Background] De Shazer, S., & Berg, I. K. (1997). "What works?" Remarks on research aspects of Solution-Focused Brief Therapy. Journal of Family Therapy, 19(2). https://doi.org/10.1111/1467-6427.00043
- [Background] De Shazer S, Berg IK, Lipchik E, Nunnally E, Molnar A, Gingerich W, Weiner-Davis M. Brief therapy: focused solution development. Fam Process. 1986 Jun;25(2):207-21. doi: 10.1111/j.1545-5300.1986.00207.x. PMID 3732502
- [Background] Erbe D, Eichert HC, Riper H, Ebert DD. Blending Face-to-Face and Internet-Based Interventions for the Treatment of Mental Disorders in Adults: Systematic Review. J Med Internet Res. 2017 Sep 15;19(9):e306. doi: 10.2196/jmir.6588. PMID 28916506
- [Background] Geschwind N, Arntz A, Bannink F, Peeters F. Positive cognitive behavior therapy in the treatment of depression: A randomized order within-subject comparison with traditional cognitive behavior therapy. Behav Res Ther. 2019 May;116:119-130. doi: 10.1016/j.brat.2019.03.005. Epub 2019 Mar 9. PMID 30897464
- [Background] Grant, A. M. (2012). Making Positive Change: A Randomized Study Comparing Solution-Focused vs. Problem-Focused Coaching Questions. Journal of Systemic Therapies, 31(2). https://doi.org/10.1521/jsyt.2012.31.2.21
- [Background] Grant, A. M., & O'Connor, S. A. (2010). The differential effects of solution-focused and problem-focused coaching questions: A pilot study with implications for practice. Industrial and Commercial Training, 42(2). https://doi.org/10.1108/00197851011026090
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Padesky CA, Mooney KA. Strengths-based cognitive-behavioural therapy: a four-step model to build resilience. Clin Psychol Psychother. 2012 Jul-Aug;19(4):283-90. doi: 10.1002/cpp.1795. Epub 2012 Jun 1. PMID 22653834
- [Background] Seligman, M. E. (2002). Positive psychology, positive prevention, and positive therapy. Handbook of positive psychology, 2(2002), 3-12.
- [Background] Seligman, M. E. (2002). Authentic happiness: Using the new positive psychology to realize your potential for lasting fulfillment. Simon and Schuster.
- [Background] Tomoiagă, C., & David, O. (2023). Is cognitive-behavioral coaching an empirically supported approach to coaching? a meta-analysis to investigate its outcomes and moderators. Journal of Rational-Emotive & Cognitive-Behavior Therapy, 41(2), 489-510. https://doi.org/10.1007/s10942-023-00498-y